CLINICAL TRIAL: NCT06319807
Title: Using Digital Health Technologies to Prevent Obesity Among Infants of Parents Receiving Nutrition Assistance Benefits.
Brief Title: GrowWell - Responsive Bottle Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00110194
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-01

CONDITIONS: Bottle Feeding
Keywords: obesity prevention; Women, Infants, and Children )WIC); infant growth
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Intervention (Experimental): Participants will receive: 1) tailored behavior change goals, 2) self-monitoring with tailored feedback, and 3) tips to foster self-efficacy and skills training around responsive feeding - provide fully automated tailored feedback, which will include theory-driven content that aims to normalize common issues and problems, provide active solutions to feeding problems and affirm positive behavior. Participants will receive daily text messages for 12 weeks. Twice a week participants will be asked to self-monitor their adherence to goals in response to a text messaging prompt and will immediately receive tailored feedback and tips.
  Interventions: Behavioral: Digital Health Intervention
- Safety Control (Active Comparator): Participants will receive tips to foster self-efficacy and skills training around infant safety. Participants will receive daily text messages for 12 weeks. Twice a week participants will be asked to self-monitor their adherence to safety goals in response to a text messaging prompt and will immediately receive tailored feedback and tips.
  Interventions: Behavioral: Safety Control

INTERVENTIONS:
Behavioral: Digital Health Intervention — Participants will receive: 1) behavior change goals, 2) self-monitoring with tailored feedback, and 3) skills training. We will use text messaging to administer the intervention pieces. At baseline, each participant will complete a series of surveys to gain background information. Throughout the study participants will report their goal adherence in response to a text messaging prompt and immediately receive tailored feedback. Text messages will be deployed daily with 2 check in messages per week; participants will receive tailored feedback based on their response.
  Arms: Digital Health Intervention
Behavioral: Safety Control — Participants will receive: 1) behavior change goals, 2) self-monitoring with tailored feedback, and 3) skills training. We will use text messaging to administer the intervention pieces. At baseline, each participant will complete a series of surveys to gain background information. Throughout the study participants will report their goal adherence in response to a text messaging prompt and immediately receive tailored feedback. Text messages will be deployed daily with 2 check in messages per week; participants will receive tailored feedback based on their response.
  Arms: Safety Control

SUMMARY:
The overall goal of this research is use digital health to augment the clinical encounter with Women, Infants, and Children (WIC) clinicians and prevent rapid infant weight gain among children living in low-income households. Intervening on weight gain during infancy offers an opportunity to influence lifelong obesity risk. Using personalized motivational messages and targeted skills-training resources, the intervention will support parents and caregivers in adopting responsive feeding strategies. Knowledge gained from this project will be used to develop a future, larger grant submission focused on developing healthy feeding and eating habits among mother-infant dyads.

DETAILED DESCRIPTION:
Assess the feasibility and acceptability of a digital intervention aimed at increasing responsive infant feeding behaviors, beginning 1 month postpartum and continuing through 3-months postpartum, among a prospective cohort of women receiving WIC benefits.

Use qualitative methods to explore barriers and facilitators to participation in a digital infant feeding intervention among women receiving WIC benefits during early postpartum

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* as a smartphone and an email address
* willing to send and receive daily text messages
* can read and write in English
* child is <=6 weeks

Exclusion Criteria:

* participating in in a different research study that, in the opinion of the investigator, would conflict or would otherwise be too problematic if the subject were to participate in this study
* planning to leave North Carolina in the next 6 months
* subjects who do not have the capacity to give legally effective consent
* any medical or congenital condition that would interfere with infant feeding or growth (ie, Down syndrome or cleft lip or palate)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Engagement - average text message completion rate | Week 12
  Engagement will be assessed by reporting the average text message completion rate over the 12-week intervention period.

SECONDARY OUTCOMES:
Satisfaction Scores - Acceptability | Week 12
  Satisfaction with the intervention content - Participants will be asked to complete satisfaction surveys upon study completion to assess the acceptability of the message perceptions about the use of digital technologies. There isn't a scale; we will report percentage responding positively to each question.
Satisfaction Scores - Frequency | Week 12
  Satisfaction with the intervention message frequency - Participants will be asked to complete satisfaction surveys upon study completion to assess the frequency of the use of digital technologies. There isn't a scale; we will report percentage responding positively to each question.
Satisfaction Scores - Timing | Week 12
  Satisfaction with the intervention message timing - Participants will be asked to complete satisfaction surveys upon study completion to assess the timing, of the use of digital technologies. There isn't a scale; we will report percentage responding positively to each question.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa C Kay, PhD, Principal Investigator — Wake Forest University Health Sciences; Sarah M Shelton, BSN, Study Director — Atrium Health Wake Forest Baptist
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT06319807/ICF_000.pdf